CLINICAL TRIAL: NCT05440981
Title: The Use of Temporarily Implanted Nitinol Device (iTind) System in Chinese Male Patients With Lower Urinary Tract Symptom Secondary to Benign Prostate Enlargement
Brief Title: Implanted Nitinol Device (iTind) System in Chinese Males With Lower Urinary Tract Symptom Secondary to BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2022.244
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporarily implanted nitinol device (iTind) group (Experimental): Subjects will undergo iTind for the treatment of male LUTS.
  Interventions: Device: iTind device

INTERVENTIONS:
Device: iTind device — Cystoscopy will be performed to assess the anatomy of the bladder and prostate. The iTind device would be inserted under visual guidance into the bladder. The device will then be deployed and under visual guidance, it will be positioned at the prostatic lumen. After confirming the position of the device, cystoscopy will be withdrawn and the position will be finished.

SUMMARY:
This is a prospective series of consecutive cases of patients undergoing iTind for the treatment of male LUTS.

DETAILED DESCRIPTION:
This is a prospective series of consecutive cases of patients undergoing iTind for the treatment of male LUTS.The procedure was carried out using perioperative antibiotic prophylaxis, according to the local culture and sensitivity profile. Patient will be discharged and readmitted 7 days for device removal under local anaesthesia transurethrally. After the device is removed and patients will be monitor for any problem in voiding or haematuria, and then discharged. Subjects will be follow-up at 3-, 6, 12- months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 50 - 80 years
* Clinically indicated for surgical treatment
* Prostate volume of 25 to 75 cc

Exclusion Criteria:

* Patients with active urinary tract infection or in retention of urine
* Patients with bleeding disorder or on anti-coagulation
* Patients with bladder pathology including bladder stone and bladder cancer
* Patients with urethral stricture
* Patients with neurogenic bladder and/or sphincter abnormalities
* Patients with previous nonpharmacological prostate treatment,
* Prostate cancer
* Fail to give informed consent

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Changes in International Prostate Symptom Score (IPSS) at 6 months after treatment score | Baseline and 6 months
  Change in total scores in International Prostate Symptom Score (ranges from 0 to 35) questionnaires.The higher score the more worse symptom.

SECONDARY OUTCOMES:
30-day complications after study intervention | at 30 days after study intervention
  The severity of AE is grade by Clavien-Dindo classification.The higher score, the more worse complication
Total score in IPSS questionnaire after study intervention | Baseline, 3 months, 6 months and 12 months
  International Prostate Symptom Score (ranges from 0 to 35) questionnaires. The higher score the more worse symptom.
International Prostate Symptom Score (IPSS) questionnaire QoL Score | Baseline, 3 months, 6 months and 12 months
  Change in quality of life assessed by International Prostate Symptom Score questionnaire (ranges from 0 to 6). The lower score the more worse QoL
Overactive bladder symptom score (OABSS) questionnaire total score | Baseline, 3 months, 6 months and 12 months
  Change in total score in Overactive Bladder Symptom Score questionnaire (ranges from 0 - 15). The higher score the more worse symptom
Pain Score | Immediately after study intervention and 1 wee after study intervention
  Post-treatment pain score ranges from 1 to 10. The higher score the more pain.
Urodynamic function assessed by uroflowmetry parameter | Baseline, 3 months, 6 months and 12 months
  Change in Maximum uroflow, post void residual

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahokehr A, Gilling PJ. Landmarks in BPH--from aetiology to medical and surgical management. Nat Rev Urol. 2014 Feb;11(2):118-22. doi: 10.1038/nrurol.2013.318. Epub 2014 Jan 21. PMID 24445912
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Amparore D, Fiori C, Valerio M, Schulman C, Giannakis I, De Cillis S, Kadner G, Porpiglia F. 3-Year results following treatment with the second generation of the temporary implantable nitinol device in men with LUTS secondary to benign prostatic obstruction. Prostate Cancer Prostatic Dis. 2021 Jun;24(2):349-357. doi: 10.1038/s41391-020-00281-5. Epub 2020 Oct 1. PMID 33005003
- [Background] Chughtai B, Elterman D, Shore N, Gittleman M, Motola J, Pike S, Hermann C, Terrens W, Kohan A, Gonzalez RR, Katz A, Schiff J, Goldfischer E, Grunberger I, Tu LM, Alshak MN, Kaminetzky J. The iTind Temporarily Implanted Nitinol Device for the Treatment of Lower Urinary Tract Symptoms Secondary to Benign Prostatic Hyperplasia: A Multicenter, Randomized, Controlled Trial. Urology. 2021 Jul;153:270-276. doi: 10.1016/j.urology.2020.12.022. Epub 2020 Dec 26. PMID 33373708